CLINICAL TRIAL: NCT05968170
Title: A Feasibility Study Using the CliniMACS® Device for T-Cell Receptor (TCR) αβ+CD3+/CD19+ Depleted Hematopoietic Stem Cells for Patients Undergoing Transplant
Brief Title: TCRαβ/CD19 Depletion of Stem Cell Grafts for Transplant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding available.
Sponsor: Neena Kapoor, M.D. (Other)
Responsible Party: Sponsor-Investigator, Neena Kapoor, M.D., Sponsor-Investigator, Children's Hospital Los Angeles
Organization: Children's Hospital Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-23-00327; NCI-2024-07368 (Registry Identifier: NCI Trial Identifier)
Record Dates: First submitted 2022-04-18; First posted 2023-08-01 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Graft Vs Host Disease; Graft-versus-host-disease; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Non-hematologic Malignancy; Hematologic Malignancy
Keywords: Reduce Graft Vs Host Disease; Transplant; Depletion of Stem Cell Grafts
MeSH Terms: conditions — Graft vs Host Disease; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Patients receiving allogeneic hematopoietic stem cell transplants (Experimental): The test product is an αβ+/CD19+ T-cell depleted stem cell product using the CliniMACS system. The test product is given intravenously over a period of time as dictated by the final volume of the infused product (5mL/kg/hour).
  The target dose of CD34+ cells is 20-40 x 10^6/kg, but a minimum of 5 x 10^6/kg is required. The target dose of TCRαβ+ T-cells and CD19+/CD20+ T-cells is ≤ 1 x 10^5/kg.
  Interventions: Device: CliniMACS® device

INTERVENTIONS:
Device: CliniMACS® device — CliniMACS TCR αβ+/CD19+ cell depletion for related or unrelated haploidentical/mismatched/matched hematopoietic stem cell transplant patients and/or high risk GVHD patients.
  Other Names: CliniMACS® CD19 reagent system; CliniMACS® depletion tubing set; CliniMACS® TCR α/β reagent system

SUMMARY:
The CliniMACS® device is FDA-approved only for one indication (CD34+ selection). Additional use of this device outside of this indication requires the use of feasibility studies.

Children, adolescents and young adults with malignant and non-malignant conditions undergoing hematopoietic stem cell transplants will have stem cells selected using alpha-beta+/CD19+ cell depletion. This is a single arm feasibility study using this processing of peripheral stem cells with alternative donor sources (haploidentical, mismatched, matched unrelated) to determine efficacy as seen by engraftment and graft-versus-host disease (GVHD).

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is recognized as an effective cure for a wide range of diagnoses including hematologic malignancies, bone marrow failure syndromes, red blood cell disorders (sickle cell, beta thalassemia), white blood cell disorders (CGD), and immune deficiency disorders. Current therapy with allogeneic HCT from HLA-matched sibling donors has shown to be a potentially curative option for children with high-risk and/or relapsed hematologic malignancies (ALL/AML) as well as primary immune deficiency disorders (PID), however only 25-30% of patients have an HLA-identical matched sibling. Alternative stem cell sources include matched unrelated donors (MUD) and unrelated cord blood (UCB), however, the likelihood of finding an unrelated match can range between 29-79% depending on the patient's ethnic background. Since 2015, the CHLA Transplant and Cellular Therapy Program has performed approximately 90 ex vivo processed haploidentical transplants. Greater than 80% of our patients belong to racial/ethnic groups with limited unrelated donor availability, relying heavily on haploidentical donors. This lack of matched stem cells represents a significant access disparity for underrepresented minorities with life-threatening hematologic or immunologic conditions to undergo a potentially curative HSCT.

The FDA approved the use of the CliniMACS CD34+ Reagent System as a Humanitarian Use Device for the prevention of GVHD in patients with acute myeloid leukemia (AML) in first complete remission undergoing allogeneic hematopoietic stem cell transplantation (HSCT) from a matched related donor. The CliniMACS CD34+ Reagent System decreases the risk of developing GVHD by efficiently removing donor T-cells from the graft prior to infusion by enriching CD34+ blood stem cells, which help to repopulate the patient's immune system. FDA approval was based on data from a phase II, single-arm, multi-center study conducted by the Blood and Marrow Transplant Clinical Trials Network that showed after an intensive myeloablative conditioning, receiving a stem cell transplant from a matched related donor processed through the CliniMACS CD34+ Reagent System as a GVHD prophylaxis led to a low incidence of chronic GVHD, about 19% at 2 years post-transplant. However, removal of all cells except CD34+ selected complicates immune recovery (delay in CD4+ cells) leading to higher rates of opportunistic viral infections and transplant-related mortality.

The use of CD34+ selected processing has facilitated approximately 42 HSCTs in combination of TCRαβ+/CD19 depletion at CHLA. The new approach to ex vivo processing utilizes negative depletion of cells thought to be responsible for the development of aGVHD, αβ TCR positive T-cells and includes simultaneous depletion of CD19+ B-cells. Since 2015, CHLA has conducted TCRαβ/CD19+ depleted HSCTs successfully on several protocols, including the ONC1401 KIR Study (IDE#16412).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (and written assent, if applicable) obtained prior to enrollment.
* Age < 21.
* Lansky Play-Performance Scale or Karnofsky Index score ≥ 60%.
* Adequate organ function (within 4 weeks of initiation of preparative regimen) as evaluated per institutional guidelines. Adequate major organ system function as demonstrated by:

  * Renal: Creatinine clearance or GFR of ≥ 60mL/min/1.73m2.
  * Hepatic: total bilirubin < 2 mg/dL (unless due to Gilbert syndrome) and ALT/AST ≤ 2.5 times the upper limit of normal.
  * Cardiac: LVEF at rest ≥ 50% or SF ≥ 27% (by MUGA or ECHO).
  * Pulmonary: DLCO, FEV1, and FVC ≥ 50% of predicted corrected for hemoglobin. For patients < 7 years of age or those unable to perform PFTs: O2 Sat ˃ 92% on room air by pulse oximetry and on no supplemental O2 at rest.
* Available donor (matched/mismatched unrelated, mismatched related, related haploidentical) who is healthy and willing to donate peripheral blood stem cells.
* Patients that have been diagnosed with graft rejection/failure or relapse may be eligible to receive a second transplant pending patient status.

Exclusion Criteria:

* Patients with HIV or uncontrolled fungal, bacterial, or viral infections.
* Patients with active CNS leukemia or any other active site of extramedullary disease at the time of enrollment.
* Recipient with HLA antibody against donor.
* Patients that are pregnant, breastfeeding or unwilling to practice birth control during participation of the study.
* Any condition that, in the opinion of the Sponsor-Investigator, would compromise the safety of the participant, prevent study participation, or interfere with the evaluation of study endpoints.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05-27 (Estimated); Primary Completion 2028-05-27 (Estimated); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3-4 acute and/or chronic GVHD at Day+100 | Day+100 post-HSCT
  Assess the cumulative incidence of severe GVHD following HSCT with TCRαβ+/CD19+ T-cell depleted grafts, as determined by the presence of Grade III-IV aGVHD and/or cGVHD by Day+100 post-HSCT.

SECONDARY OUTCOMES:
Incidence of engraftment at Day+30. | Day+30 post-HSCT
  Assess the efficacy of TCRαβ+/CD19+ T-cell depleted HSCTs as measured by the engraftment of donor cells by Day+30 post-HSCT.
Incidence of transplant-related mortality at 1-year post-HSCT. | 1-Year post-HSCT
  Assess the efficacy of TCRαβ+/CD19+ T-cell depleted HSCTs as measured by the incidence of transplant-related mortality at 1-year post-HSCT.
Incidence of T-cell reconstitution at Day+180 (CD4+ T-cell count > 200 and proliferation to PHA > 50% control). | Day+180 post-HSCT
  Assess the immune reconstitution following TCRαβ+/CD19+ T-cell depleted HSCTs as measured by the presence of expanded T-cell numbers and function at Day+180 post-HSCT(CD4+ T-cell count > 200 and proliferation to PHA > 50% control).

OTHER OUTCOMES:
Incidence of microbial contamination of the infused cells product leading to possible infection in the recipient (i.e., antibiotics needed for > 48 hours). | Day+30
  Assess the risk of microbial contamination in TCRαβ+/CD19+ T-cell depleted products from the CliniMACS® device.

CONTACTS AND LOCATIONS:
Overall Officials: Neena Kapoor, MD, Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available internally to other sub-investigators that have expressed interest. Data that will be shared must go through the Sponsor-Investigator and will be redacted (if not already done) prior to receiving the data so that no identifying information is present.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available upon request by submitting criteria of interest. The Sponsor-Investigator will provide a copy of the data. The copy will be indefinitely available to the interested party.
Access Criteria: Data will be made available upon request by submitting criteria of interest. A copy of the redacted data will be given. No other party will have access to the database at any time outside of the Sponsor-Investigator and data management/CRC team.

REFERENCES:
- [Background] Oliansky DM, Rizzo JD, Aplan PD, Arceci RJ, Leone L, Ravindranath Y, Sanders JE, Smith FO 3rd, Wilmot F, McCarthy PL Jr, Hahn T. The role of cytotoxic therapy with hematopoietic stem cell transplantation in the therapy of acute myeloid leukemia in children: an evidence-based review. Biol Blood Marrow Transplant. 2007 Jan;13(1):1-25. doi: 10.1016/j.bbmt.2006.10.024. PMID 17222748
- [Background] Oliansky DM, Camitta B, Gaynon P, Nieder ML, Parsons SK, Pulsipher MA, Dillon H, Ratko TA, Wall D, McCarthy PL Jr, Hahn T; American Society for Blood and Marrow Transplantation. Role of cytotoxic therapy with hematopoietic stem cell transplantation in the treatment of pediatric acute lymphoblastic leukemia: update of the 2005 evidence-based review. Biol Blood Marrow Transplant. 2012 Apr;18(4):505-22. doi: 10.1016/j.bbmt.2011.12.585. Epub 2011 Dec 29. PMID 22209888
- [Background] Leung W, Campana D, Yang J, Pei D, Coustan-Smith E, Gan K, Rubnitz JE, Sandlund JT, Ribeiro RC, Srinivasan A, Hartford C, Triplett BM, Dallas M, Pillai A, Handgretinger R, Laver JH, Pui CH. High success rate of hematopoietic cell transplantation regardless of donor source in children with very high-risk leukemia. Blood. 2011 Jul 14;118(2):223-30. doi: 10.1182/blood-2011-01-333070. Epub 2011 May 25. PMID 21613256
- [Background] Fuchs EJ. Haploidentical transplantation for hematologic malignancies: where do we stand? Hematology Am Soc Hematol Educ Program. 2012;2012:230-6. doi: 10.1182/asheducation-2012.1.230. PMID 23233586
- [Background] Zeidan AM, Forde PM, Symons H, Chen A, Smith BD, Pratz K, Carraway H, Gladstone DE, Fuchs EJ, Luznik L, Jones RJ, Bolanos-Meade J. HLA-haploidentical donor lymphocyte infusions for patients with relapsed hematologic malignancies after related HLA-haploidentical bone marrow transplantation. Biol Blood Marrow Transplant. 2014 Mar;20(3):314-8. doi: 10.1016/j.bbmt.2013.11.020. Epub 2013 Dec 1. PMID 24296490
- [Background] Food and Drug Administration, HHS. Eligibility determination for donors of human cells, tissues, and cellular and tissue-based products. Final rule. Fed Regist. 2004 May 25;69(101):29785-834. PMID 15160713
- [Background] Food and Drug Administration, HHS. Current good tissue practice for human cell, tissue, and cellular and tissue-based product establishments; inspection and enforcement. Final rule. Fed Regist. 2004 Nov 24;69(226):68611-88. PMID 15562555
- [Background] Abdelhakim H, Abdel-Azim H, Saad A. Role of alphabeta T Cell Depletion in Prevention of Graft versus Host Disease. Biomedicines. 2017 Jun 26;5(3):35. doi: 10.3390/biomedicines5030035. PMID 28672883
- [Background] Radestad E, Sundin M, Torlen J, Thunberg S, Onfelt B, Ljungman P, Watz E, Mattsson J, Uhlin M. Individualization of Hematopoietic Stem Cell Transplantation Using Alpha/Beta T-Cell Depletion. Front Immunol. 2019 Feb 11;10:189. doi: 10.3389/fimmu.2019.00189. eCollection 2019. PMID 30804948
- [Background] Ciurea SO, Bayraktar UD. "No donor"? Consider a haploidentical transplant. Blood Rev. 2015 Mar;29(2):63-70. doi: 10.1016/j.blre.2014.09.009. Epub 2014 Sep 30. PMID 25307958
- [Background] Gournay V, Dumas G, Lavillegrand JR, Hariri G, Urbina T, Baudel JL, Ait-Oufella H, Maury E, Brissot E, Legrand O, Malard F, Mohty M, Guidet B, Dulery R, Bige N. Outcome of allogeneic hematopoietic stem cell transplant recipients admitted to the intensive care unit with a focus on haploidentical graft and sequential conditioning regimen: results of a retrospective study. Ann Hematol. 2021 Nov;100(11):2787-2797. doi: 10.1007/s00277-021-04640-7. Epub 2021 Sep 3. PMID 34476574
- [Background] Giardino S, Bagnasco F, Falco M, Miano M, Pierri F, Risso M, Terranova P, Di Martino D, Massaccesi E, Ricci M, Chianucci B, Dell'Orso G, Sabatini F, Podesta M, Lanino E, Faraci M. Haploidentical Stem Cell Transplantation After TCR-alphabeta+ and CD19+ Cells Depletion In Children With Congenital Non-Malignant Disease. Transplant Cell Ther. 2022 Jul;28(7):394.e1-394.e9. doi: 10.1016/j.jtct.2022.04.002. Epub 2022 Apr 8. PMID 35405368
- [Background] Arnold DE, MacMath D, Seif AE, Heimall JR, Wang Y, Monos D, Grupp SA, Bunin NJ. Immune Reconstitution Following TCRalphabeta/CD19-Depleted Hematopoietic Cell Transplantation for Hematologic Malignancy in Pediatric Patients. Transplant Cell Ther. 2021 Feb;27(2):169.e1-169.e9. doi: 10.1016/j.jtct.2020.10.006. Epub 2020 Dec 10. PMID 33830028
- [Background] Mitchell R, Cole T, Shaw PJ, Mechinaud F, O'Brien T, Fraser C. TCR alpha+ beta+ /CD19+ cell-depleted hematopoietic stem cell transplantation for pediatric patients. Pediatr Transplant. 2019 Sep;23(6):e13517. doi: 10.1111/petr.13517. Epub 2019 Jul 4. PMID 31271477
- [Background] Bethge WA, Eyrich M, Mielke S, Meisel R, Niederwieser D, Schlegel PG, Schulz A, Greil J, Bunjes D, Brecht A, Kuball J, Schumm M, Vucinic V, Wiesneth M, Bonig H, Westinga K, Biedermann S, Holtkamp S, Karitzky S, Malchow M, Siewert C, Handgretinger R, Lang P. Results of a multicenter phase I/II trial of TCRalphabeta and CD19-depleted haploidentical hematopoietic stem cell transplantation for adult and pediatric patients. Bone Marrow Transplant. 2022 Mar;57(3):423-430. doi: 10.1038/s41409-021-01551-z. Epub 2021 Dec 24. PMID 34952929